CLINICAL TRIAL: NCT01086579
Title: Balloon Elution and Late Loss Optimization (BELLO) Study: A Multicentre Randomized Study of the IN.PACT Falcon™ Paclitaxel Drug-eluting Balloon to Reduce Restenosis in Small Coronary Vessels
Brief Title: Balloon Elution and Late Loss Optimization (BELLO) Study
Acronym: BELLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Evidence per Attività e Ricerche Cardiovascolari ONLUS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BELLO
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Artery Disease
Keywords: paclitaxel PTCA drug-eluting balloon; provisional spot stenting; coronary artery disease; Late Lumen Loss; Minimal lumen diameter; coronary artery disease in a small vessel
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (IN.PACT Falcon Drug Eluting Balloon) (Experimental): IN.PACT Falcon™ paclitaxel drug-eluting balloon (DEB) dilatation and provisional spot bare metal stenting (Bare Metal Stent).
  Interventions: Device: IN.PACT Falcon paclitaxel eluting balloon (Drug eluting balloon)
- Control Arm PES (Active Comparator): Control Arm: paclitaxel-eluting stent (PES) implantation as per standard practice.
  Interventions: Device: Taxus (Paclitaxel eluting stent)

INTERVENTIONS:
Device: IN.PACT Falcon paclitaxel eluting balloon (Drug eluting balloon) — Coronary Artery Bypass Graft (CABG)
  Other Names: IN.PACT Falcon paclitaxel eluting balloon
  Arms: Treatment Arm (IN.PACT Falcon Drug Eluting Balloon)
Device: Taxus (Paclitaxel eluting stent) — Percutaneous transluminal coronary angioplasty (PTCA) with stent
  Arms: Control Arm PES

SUMMARY:
Prospective multicentre randomized (1:1) investigator initiated study, in which consecutive patients undergoing percutaneous revascularization of small coronary vessels will be assigned to one of the two study arms:

1. Treatment Arm: IN.PACT Falcon™ paclitaxel drug-eluting balloon (DEB) dilatation and provisional spot bare-metal stenting (BMS).
2. Control Arm: paclitaxel-eluting stent (PES) implantation as per standard practice.

Eligible subjects with coronary artery disease in a small vessel (reference diameter<2.8mm) will be consecutively screened and enrolled based on the inclusion and exclusion criteria

The objective of the study is to assess the non-inferiority of the DEB to the PES as regards to primary endpoint of mean late lumen loss (LLL) at 6 months, defined as the difference between postprocedural minimum luminal (MLD) diameter and follow-up MLD, as assessed by quantitative coronary angiography and is based on the following assumptions:

1. The means of LLL in the 2 groups are precisely equal
2. A standard deviation in LLL of 0.5mm in both groups as demonstrated in the ISAR-SMART 3 and PEPCAD II trials
3. A non-inferiority margin of 0.25mm between groups is clinically unimportant

Based on these assumptions:

1. Null hypothesis (N0): mean LLL in DEB group is ≥0.25mm than that in the PES group (i.e. PES is superior to DEB)
2. Alternative hypothesis 1 (H1): mean LLL between DEB and PES is <0.25mm (i.e. DEB is non-inferior to PES)
3. Alternative hypothesis 2 (H2): mean LLL between DEB and PES <0 (i.e. DEB is superior to PES) Based on the above calculations, a sample size of 77 patients will be required in each group to show non-inferiority of DEB vs. PES with an α error of 0.025 (one-sided Z test) and a power of 80%. To account for a 20% rate of withdrawal, lost to follow-up or not presenting for follow-up angiography, a total of 182 patients (91 in each group) will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Patient providing written informed consent.
* Patients with stable angina pectoris (Canadian Cardiovascular Society [CCS] 1, 2 3) or unstable angina pectoris with documented ischemia (CCS 4, Braunwald Class IB-C, IIB-C or IIIB-C), or patients with documented silent ischemia.
* Patients who are eligible for coronary revascularization (angioplasty and/or CABG).
* Female patients with child bearing potential must have a negative pregnancy test within one week before treatment and must use adequate contraception.

Angiographic Inclusion Criteria:

* Native coronary artery.
* De novo lesion.
* Reference vessel diameter < 2.8mm by visual estimate.
* Target lesion with a visually estimated stenosis >50%.
* Target lesion length < 25mm by visual estimate.
* A maximum of 2 epicardial vessels requiring revascularization.
* A maximum of 2 target lesions can be included (In the case of treatment of more than one lesion, the treatment selected will remain the same).

Exclusion Criteria:

* Patients unable to give informed consent.
* Patients enrolled in another study with any investigational drug or device within the past 30 days.
* Patients scheduled for a major surgical intervention within 6 months of enrolment in the study.
* Patients with acute (< 24h) or recent (≤ 48 hours) myocardial infarction.
* Patients with a contraindication to an emergency coronary bypass surgery.
* Any individual who may refuse a blood transfusion.
* Patients with serum creatinine >2.0mg/dL or >180umol/L.
* Patients with severe congestive heart failure.
* Patients who had a cerebral stroke <6 months prior to the Index Procedure.
* EF (Ejection Fraction) < 30%.
* Patients with any known allergy, hypersensitivity or intolerance to acetylsalicylic acid (ASA), Clopidogrel or Ticlopidine, Paclitaxel.
* Any known allergy to contrast medium that cannot be pre-treated.

Angiographic exclusion criteria:

* >2 epicardial vessels requiring revascularization.
* Target lesion distance from the ostium of left anterior descending coronary artery (LAD)/left circumflex coronary artery (LCX)/right coronary artery (RCA) is < 5 mm.
* Target lesion is located in either a venous or arterial graft.
* Target vessel contains a previously implanted stent.
* Angiographic evidence of thrombus at the target site.
* Chronic total occlusions.
* Restenotic lesions.
* Bifurcation lesions which the operator decides a 2-stent technique as intention-to-treat is required OR bifurcations with side branches ≥ 2.5mm.
* Failure to successfully treat non-target lesions within the target vessel (non-target lesions must be treated prior the target lesion).
* Greater than 2 non-target lesions treated during the index procedure.
* Previous Percutaneous Coronary Intervention (PCI) within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Late Lumen Loss (LLL) at 6 months follow-up defined as the difference between postprocedural minimum luminal diameter and follow-up minimum luminal diameter, as assessed by quantitative coronary angiography | 6 Month

SECONDARY OUTCOMES:
Device Success: ability of the Investigational Device to be delivered, dilate, and be retrieved from the target lesion. | day 1
Procedural Success: defined as Device Success without the occurrence of Major Adverse Cardiac Events (MACE) during the index hospitalization | day 1
MACE rate through 30 days, 6 months,1, 2, 3 years post index procedure | 30 days, 6 months,1, 2, 3 years
Target Lesion Revascularization (TLR) at 6 months,1, 2, 3 years post index procedure | 6 months,1, 2, 3 years
Target Vessel Revascularization (TVR) at 6 months,1, 2, 3 years post index procedure | 6 months,1, 2, 3 years
Target vessel failure (TVF), defined as cardiac death, Myocardial Infarction (MI) or TVR at 1 year | 1 Year
Binary Restenosis rate at 6 months follow-up | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, Dr., Principal Investigator — IRCCS Fondazione Centro S.Raffaele del Monte Tabor; Corrado Tamburino, Prof., Principal Investigator — Presidio Ospedaliero Ferrarotto di Catania; Patrizia Presbitero, Prof, Principal Investigator — Istituto Clinico Humanitas di Rozzano (MI); Alberta Pangrazi, Dr., Principal Investigator — Azienda Ospedaliera Ospedali Riuniti Umberto I-G.M.Lancisi-G.Salesi di Ancona; Roberto Violini, Dr., Principal Investigator — Azienda Ospedaliera San Camillo Forlanini di Roma; Francesca Buffoli, Dr., Principal Investigator — Ospedale "C.Poma" di Mantova; Maurizio Tespili, Dr., Principal Investigator — Azienda Ospedaliera "Bolognini" di Seriate; Fausto Castriota, Dr., Principal Investigator — Citta' di Lecce Hospital di Lecce; Alberto Cremonesi, Dr., Principal Investigator — Villa Maria Cecilia Hospital di Cotignola; Antonio Micari, Dr., Principal Investigator — Villa Maria Eleonora Hospital di Palermo; Alfredo Marchese, Dr., Principal Investigator — Casa di Cura "AntheaHospital" di Bari; Fabrizio Tomai, Dr., Principal Investigator — European Hospital di Roma; Massimo Margheri, Dr., Principal Investigator — Ospedale S.Maria delle Croci AUSL di Ravenna; Alberto Menozzi, Dr., Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- Irccs Fondazione Centro S.Raffaele Del Monte Tabor, Milan, MI, Italy

REFERENCES:
- [Derived] Latib A, Colombo A, Castriota F, Micari A, Cremonesi A, De Felice F, Marchese A, Tespili M, Presbitero P, Sgueglia GA, Buffoli F, Tamburino C, Varbella F, Menozzi A. A randomized multicenter study comparing a paclitaxel drug-eluting balloon with a paclitaxel-eluting stent in small coronary vessels: the BELLO (Balloon Elution and Late Loss Optimization) study. J Am Coll Cardiol. 2012 Dec 18;60(24):2473-80. doi: 10.1016/j.jacc.2012.09.020. Epub 2012 Nov 14. PMID 23158530